CLINICAL TRIAL: NCT04306250
Title: Comparison of Posterior and Anterior Approach to Sacrospinous Ligament Apical Fixation - Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Meirav Braverman, medical doctor, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 145-19
Record Dates: First submitted 2020-02-24; First posted 2020-03-12 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Organ Prolapse; Surgical Procedure, Unspecified
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- anterior approach for apical fixation to the SSL (Experimental): In this group the apical fixation will be done using the anterior access, ie dissection through the anterior vaginal wall.
  Interventions: Procedure: Apical prolapse fixation - anterior access
- posterior approach for apical fixation to the SSL (Active Comparator): In this group the apical fixation will be done using the posterior access, ie fixation through the vaginal posterior wall.
  Interventions: Procedure: Apical prolapse fixation - posterior access

INTERVENTIONS:
Procedure: Apical prolapse fixation - anterior access — The surgery is done in anterior access
  Arms: anterior approach for apical fixation to the SSL
Procedure: Apical prolapse fixation - posterior access — The surgery is done in posterior access
  Arms: posterior approach for apical fixation to the SSL

SUMMARY:
Pelvic organ prolapse (POP) is a common problem among women. Apical prolapse (AP) is a prolapse of the uterus, or vaginal cuff, in women post hysterectomy.

Apical fixation to the sacrospinous ligament (SSLF) was first introduced in 1968 by K.RICHTER. .In a large review study, the subjective cure rate after SSLF ranged from 70 to 98%, while objective cure rate was 67-97%.

The success rates of SSLF in a randomized study comparing SSLF to uterosacral ligament fixation after two years were 63.1%. In women with combined apical and anterior wall prolapse, SSLF can be performed in two ways: anterior access through the anterior vaginal wall or posterior approach through the posterior vaginal wall.

A retrospective comparison of the two methods was performed, demonstrating some efficacy to the anterior approach over the posterior approach mainly in respect to the vaginal length.

From the literature review to date, no comparisons were made between the methods in a randomized controlled trial.

Objective: To compare the success rates between two approaches (anterior and posterior) for SSLF

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a common problem among women and its incidence is rising due to population aging. Approximately 11-19% of women will undergo surgery for pelvic organ prolapse (POP) or urinary incontinence during their lifetime and approximately 30% will need repeat surgery during their lifetime .Apical prolapse (AP) is a prolapse of the uterus, or vaginal cuff, in women post hysterectomy. The severity of the prolapsed organ can be graded according to the POP-Q classification .There are several approaches to apical fixation, some of which are done vaginally and include fixation by sutures to the uterosacral ligament (USLF) or the sacrospinous ligament (SSLF). A mesh can be used for ligament fixation as well. The abdominal approach is also an option, the sacro-colpo-pexy fixation using a Y mesh. Apical fixation to the SSL was first introduced in 1968 by K.RICHTER. medical devices such as the Capio that assist in performing SSLF were also developed with ease.

In a review article that included 2,390 women undergoing SSLF subjective cure rate ranged from 70 to 98%, while objective cure rate was 67-97% .Such fixation in combination with posterior or anterior wall repair, especially after hysterectomy, showed a 94% objective cure rate at 7-year postoperative follow-up. A randomized study (The "OPTIMAL randomised trial") comparing SSLF with USLF found no preference for either method. Success rates were measured according to three criteria - 1) no significant vaginal dome or one of the vaginal walls 2) no vaginal bulge symptoms 3) no need for repeated surgery within two years of the original surgery. According to this study, the success rates of SSLF after two years were 63.1%.

Among women with anterior vaginal wall prolapse and AP, SSLF can be performed in two ways: anterior access, ie dissection through the anterior wall of the vagina or fixation through the posterior wall of the vagina. A retrospective comparison of the two methods was performed, demonstrating some efficacy in anterior approach in terms of vaginal length and postoperative apical fixation with less reference to healing rates or impact on the anterior compartment, compared with a posterior approach.

From the literature review to date, no comparisons were made between the methods in a randomized controlled trial.

Objective: To compare the success rates of two approaches (anterior and posterior) for SSLF

ELIGIBILITY:
Inclusion Criteria:

* Women with grade 2 or above apical prolapse, according to POP Q, combined with Grade II or above of anterior wall prolapse.
* Women who suffer from symptomatic POP and care for a surgical treatment

Exclusion Criteria:

* Women with a contra-indication for surgical treatment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 280 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compound cure rate | 6-month (and will be further followed yearly until 2 years of total follow up)
  A compound cure rate is composite outcome used to measure the success rate of a surgery designed to repair pelvic organ prolapse. Surgery will be considered successful based on each of the following criteria at the 6-month follow-up (and will be further followed yearly until 2 years of total follow up):
  A. Lack of apical and anterior wall prolapse beyond stage 1 (POP-Q stage<=1) b. Subjective success- a negative response ("no" or not at all to the question, "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?" (Question 3 on the PFDI-20 questionnaire), (score <2).
  c. No re-treatment (surgical/ non-surgical) for index compartment

SECONDARY OUTCOMES:
Duration of surgery | From the time of the first cut of the surgery to the time the surgery ends (as documented in the surgery report), up to 240 minutes
  Duration of surgery in minutes
Change in hemoglobin level from pre-operation level to post-operative level in g/dl units | Hb level will be measured up to 1 month before the surgery and at the 24 hours after surgery. Further examinations will be taken if there is clinical suspicious for bleeding, up to the day of discharge)
  to assess the difference in Hb level before and after the surgery
Intraoperative complications | Any complication the occured during the duration of the surgery
  Any documented event of perforation of adjacent organs such as bladder, ureter, intestine or blood vessel injury that occured during the surgery
Peri-operative complications | Any complications that occured from the end of the surgery until the first check-up visit (6 weeks after rthe surgery)
  Any event of fever / abnormal discharge / abscess / contaminated hematoma/ need for blood transfusion
Maximal pain score | Maximal pain level during the 6 weeks after the surgery
  To assess a patient's pain level, the investigators will use visual analog scale (VAS)- scale for patient self-reporting of pain. 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain, 7-10 represents severe pain).
  the investigators will assess the maximum pain level during the 6 weeks after the surgery
Change in PFDI-20 score | 6, 12 and 24 months post the operation
  Mean scores and change from baseline of PFDI-20 score at 6 and 12, 24 months. To evaluate prolapse, urinary and bowel function(PFDI-20).
Patient global impression of improvement from surgery | 6, 12 and 24 months post the operation
  Mean scores of PGI-I at 6 and 12, 24 months. To evaluate patient satisfaction from the surgery.
Cure rate at 12 months post-operation | 12 months post the operation
  A compound cure rate is composite outcome used to measure the success rate of a surgery designed to repair pelvic organ prolapse. Surgery will be considered successful based on each of the following criteria at the 12-month follow-up :
  A. Lack of apical and anterior wall prolapse beyond stage 1 (POP-Q stage<=1) b. Subjective success- a negative response ("no" or not at all to the question, "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?" (Question 3 on the PFDI-20 questionnaire), (score <2).
  c. No re-treatment (surgical/ non-surgical) for index compartment
Cure rate at 24 months post-operation | 24 months post the operation
  A compound cure rate is composite outcome used to measure the success rate of a surgery designed to repair pelvic organ prolapse. Surgery will be considered successful based on each of the following criteria at the 24-month follow-up :
  A. Lack of apical and anterior wall prolapse beyond stage 1 (POP-Q stage<=1) b. Subjective success- a negative response ("no" or not at all to the question, "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?" (Question 3 on the PFDI-20 questionnaire), (score <2).
  c. No re-treatment (surgical/ non-surgical) for index compartment
long term complications | 6, 12 and 24 months post the operation
  Incidence of new-onset dyspareunia; de-novo urinary or bowel problems; re-operation for prolapse in the index compartment; de-novo pelvic pain.

CONTACTS AND LOCATIONS:
Overall Officials: meirav breverman, MD, Principal Investigator — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel